CLINICAL TRIAL: NCT01826357
Title: Cluster Analysis of the Risk of Metabolic Syndrome in Women for Reproductive Age.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Ming-I Hsu, Taipei Medical University WanFang Hospital, Taipei Medical University WanFang Hospital
Other Study IDs: Hsu2013-TMU-JIRB 201302002
Record Dates: First submitted 2013-04-03; First posted 2013-04-08 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Metabolic Cardiovascular Syndrome
Keywords: metabolic syndrome; cluster analysis; PCOS
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The metabolic syndrome (MetS) is a cluster of clinical indices that signals increased risk for cardiovascular disease and Type 2 diabetes. Women with polycystic ovary syndrome (PCOS) were associated with MetS and insulin resistance. Cluster analysis was a useful tool for identifying groups of women sharing similar metabolic risk factor patterns. Oligomenorrhea, hyperandrogenism and polycystic ovary morphology were the three major components of PCOS. Obesity is a main risk factor in metabolic syndrome. the investigators are interesting to evaluate the relationship between risk of metabolic syndrome and their clinical and/or biochemical characteristics in women with reproductive age.

Design: Retrospective study; medical records reviewed. Participants and setting: The investigators retrospectively reviewed the medical records of female patients who visited our Reproductive Endocrinology Clinic from Jan. 1, 2009 to Jun. 31, 2012.

DETAILED DESCRIPTION:
Definitions of the metabolic syndrome based on arbitrary cutoff points for several quantitative variables, where each variable is related linearly to cardiovascular risk. Even consensual definitions differ between international authorities and continue to change. Moreover, such cutoff s should be gender and ethic difference. Cluster analysis is a statistical method base on algorithms, which seek to minimize within-group variation and maximize between-group variation for the clustering variables. This technique is suitable for defining groups, reflecting the natural structure of data without relying on inappropriate arbitrary cutoffs. We conduct this retrospective study to review the medical records of female patients who visited our Reproductive Endocrinology Clinic from Jan. 1, 2009 to Dec. 31, 2012. Cluster analysis was performed in our studied cases to evaluate the correlation between clinical/biochemical characteristic and risk of metabolic risk in women with reproductive age.

ELIGIBILITY:
Inclusion Criteria:

Women had been fulfilled with whole anthropometric measurements, clinic and biochemical survey about cardiovascular study.

Exclusion Criteria:

1. women who had been diagnosed with malignant tumor, Asherman's syndrome, Mullerian agenesis, and chromosomal anomalies;
2. women who had had menarche less than 1 years before evaluation or who were older than 49;
3. women who received hormones or drugs for major medical diseases within three months of blood sampling.

Ages: 13 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women had been fulfilled with whole anthropometric measurements, clinic and biochemical survey about cardiovascular study.
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
metabolic syndrome | Retrospectively reviewed the patients who visited Reproductive Endocrinology Clinic from Jan. 1, 2009 to Jun. 31, 2012.
  We conduct this retrospective study by using cluster analysis, to investigate the relationship between metabolic complications and biochemical/clinical characteristics of endocrinologic dysfunction in women with reproductive age.

CONTACTS AND LOCATIONS:
Overall Officials: Ming I Hsu, MD, Principal Investigator — WanFang Medical Center at Taipei Medical University
Locations (1):
- WanFang Medical Center at Taipei Medical University, Taipei, Taiwan, Taiwan

REFERENCES:
- [Derived] Tzeng CR, Chang YC, Chang YC, Wang CW, Chen CH, Hsu MI. Cluster analysis of cardiovascular and metabolic risk factors in women of reproductive age. Fertil Steril. 2014 May;101(5):1404-10. doi: 10.1016/j.fertnstert.2014.01.023. Epub 2014 Feb 15. PMID 24534286